CLINICAL TRIAL: NCT07173257
Title: Patient Reported Outcomes Measures in Patients Undergoing Pancreatic Resections
Brief Title: PROMs After Pancreatectomy
Acronym: PERSPECTIVE
Status: Recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: Mayo Clinic - Scottsdale/Phoenix, Arizona (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00002020
Record Dates: First submitted 2025-03-27; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pancreas Neoplasms; Pancreatitis; Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The standard of care for a patient with resectable pancreatic is to perform pancreatic resection which, even in the modern era is associated with significant complications and impact on quality of life, often in the setting of poor survival even in the best scenario. Currently, there is a lack of data on patient quality of life after such procedures, how quality of life changes throughout the course of care, and whether patients who undergo these procedures are satisfied with their decision. This research is aimed to understand the impact of pancreatic surgery on patients' quality of life, how that impact changes over time, and patient satisfaction (or regret) with their decisions. This work will help improve the pre-operative conversation to help patients decide whether undergoing a pancreatic resection aligns with their post-operative goals of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old who undergo pancreatic resection for any indication of any race, gender, or ethnicity who are fluent in English

Exclusion Criteria:

* <18 years old
* Deemed not to have capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen at Hepato-Pancreato-Biliary Surgery Clinics for pancreatic resections will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Quality of Life Measured by EORTC QLQ-C30 Scale up to 24 Months Post-Operatively | Baseline, Immediately Post-Op, 3, 6, 12, 18, and 24 months after surgery
  The EORTC QLQ-C30 is a validated 30-item questionnaire assessing cancer-specific quality of life. The Global Health Status/QoL scale ranges from 0 to 100, with higher scores representing better quality of life.
  Unit of Measure: points Metric: Mean change from baseline Aggregation Method: Mean (SD) across participants
Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Pancreatic Cancer Module (EORTC QLQ-PAN26) Subscale Scores up to 24 Months Post-Operatively | Baseline, Immediately Post-op, 3, 6, 12, 18, and 24 months after surgery
  The EORTC QLQ-PAN26 is a 26-item, disease-specific questionnaire designed for patients with pancreatic cancer. It is used alongside the core EORTC QLQ-C30. PAN26 assesses multiple domains, including pancreatic pain, digestive symptoms, altered bowel habits, hepatic symptoms, and emotional effects. Each subscale is linearly transformed to a score from 0 to 100.
  For symptom subscales, higher scores = worse symptoms. For functioning domains, higher scores = greater impairment.
  Unit of Measure: points (0-100) per subscale Metric: mean change from baseline Aggregation: mean (SD) across participants

SECONDARY OUTCOMES:
Change from Baseline in Social Functioning (PROMIS) up to 24 Months Post-Operatively | Baseline, Immediately Post-Op, 3, 6, 12, 18, and 24 months after surgery
  PROMIS Social Isolation 8a Short Form T-score (higher = more isolation), change from baseline
Change from Baseline in Emotional Functioning (PROMIS) up to 24 Months Post-Operatively | Baseline, Immediately Post-Op, 3, 6, 12, 18, and 24 months after surgery
  PROMIS Depression 4a Short Form T-score (mean 50, SD 10; higher = more depressive symptoms), change from baseline up to 24 months post-operatively
Change from Baseline in Shared Decision-Making up to 24 Months Post-Operatively | Baseline, Immediately Post-Op, 3, 6, 12, 18, and 24 months after surgery
  Change from Baseline in Shared Decision Making Questionnaire (SDM-Q-9) Score (0-100; higher = better) up to 24 months post-operatively
  Unit: points Metric: mean change from baseline Aggregation: mean (SD)
Change from Baseline in Grit Scale (Duckworth 12-item) Total Score up to 12 Months Post-Operatively | Baseline, 6, and 12 months after surgery
  The Grit Scale is a 12-item validated self-report questionnaire that measures perseverance of effort and consistency of interests. Each item is scored from 1 ("Not at all like me") to 5 ("Very much like me"). Total scores are averaged, yielding a range of 1 to 5, with higher scores indicating greater grit.
  Unit of Measure: points (1-5) Metric: mean change from baseline Aggregation: mean (SD) across participants
Change from Baseline in Brief Resilience Scale (BRS) Score up to 24 Months Post-Operatively | Baseline, Immediately Post-Op, 3, 6, 12, and 24 months after surgery
  The Brief Resilience Scale (BRS) is a validated 6-item self-report measure assessing an individual's ability to "bounce back" from stressful events. Items are rated on a 5-point Likert scale: 1 = Strongly Disagree to 5 = Strongly Agree. After reverse-coding negatively worded items (Items 2, 4, 6), the mean of the six items is computed, yielding a score from 1.00 to 5.00: higher values reflect greater resilience.
  Unit of Measure: points (mean score) Metric: mean change from baseline Aggregation: mean (SD) across participants
Change from Baseline in COST-FACIT (Comprehensive Score for Financial Toxicity) Score up to 24 Months Post-Operatively | Baseline, Immediately Post-op, 3, 6, 12, 18, and 24 months after surgery
  The Comprehensive Score for Financial Toxicity (COST-FACIT) is an 11-item validated questionnaire that assesses the financial distress related to medical treatment. Scores range from 0 to 44, with lower scores indicating greater financial toxicity and higher scores indicating better financial well-being.
  Unit of Measure: points (0-44) Metric: mean change from baseline Aggregation: mean (SD) across participants
Change in Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF) Total Score up to 24 Months Post-Operatively | Immediately Post-op, 3, 6, 12, 18, and 24 months after surgery
  The Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF) is a 9-item validated self-report measure assessing concerns about cancer recurrence. Each item is scored on a 5-point Likert scale, yielding a total score between 0 and 36. Higher scores indicate greater fear of recurrence.
  Unit of Measure: points (0-36) Metric: mean change from baseline Aggregation: mean (SD) across participants
Change in Patient Decision Regret Scale (Brehaut et al., 2003) Total Score up to 24 Months Post-Operatively | Immediately Post-Op, 3, 6, 12, 18, and 24 months after surgery
  The Decision Regret Scale (Brehaut et al., 2003) is a validated 5-item questionnaire that assesses regret after health care decisions. Each item is scored on a 5-point Likert scale and transformed to a total score from 0 (no regret) to 100 (high regret), with higher scores reflecting greater regret.
  Units: Points (0-100) Metric: mean change from immediately post-op Aggregation: Mean (SD)
Change in Surgeon Decision Regret Scale (Brehaut et al., 2003) Total Score up to 12 Months Post-Operatively | Immediately Post-Op, 3, and 12 months after surgery
  The Decision Regret Scale (Brehaut et al., 2003) is a validated 5-item questionnaire that assesses regret after health care decisions. Each item is scored on a 5-point Likert scale and transformed to a total score from 0 (no regret) to 100 (high regret), with higher scores reflecting greater regret.
  Units: Points (0-100) Metric: mean change from immediately post-op Aggregation: Mean (SD)
Change from Baseline in Neuropathy Symptom Scores Using NCI PRO-CTCAE® Custom Item Subset up to 24 Months Post-Operatively | Baseline, 3, 6, 12, 18, and 24 months after surgery
  Neuropathy symptoms will be assessed using a custom subset of items from the U.S. National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®) v1.0 Item Library. Items address neuropathy-related domains such as numbness, tingling, pain, and interference with daily activities. Each item is scored on a 5-point Likert scale (0 = None, 4 = Very severe / Almost always / Very much). Scores can be analyzed individually or averaged per domain. Higher scores indicate greater symptom severity, frequency, or interference.
  Unit of Measure: points (0-4 per item) Metric: mean change from baseline Aggregation: mean (SD) across participants; frequency distribution of severity levels

OTHER OUTCOMES:
Themes Identified from Semi-Structured Patient Interviews on Decision-Making and Quality of Life up to 24 Months Post-Operatively | Within 24 months after surgery
  A subset of participants will be invited to complete semi-structured qualitative interviews exploring decision regret, satisfaction with the surgical decision-making process, and factors influencing post-operative quality of life. Interviews will be transcribed verbatim and analyzed using thematic analysis. Recruitment will continue until thematic saturation is achieved.
  Unit of Measure: qualitative themes (categories) Metric: number and type of themes identified; frequency of occurrence across participants Aggregation Method: descriptive summary of themes across participants

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - The University of Arizona, Tucson, Arizona